CLINICAL TRIAL: NCT04491786
Title: Department of Anaesthesiology
Brief Title: The Efficacy of Postoperative Analgesia of Gabapentin Plus Nefopam in the Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GiaDinhPH
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-01

CONDITIONS: Spinal Fusion
Keywords: Gabapentin; Nefopam; Spinal surgery; Postoperative analgesia
MeSH Terms: interventions — Gabapentin; Nefopam

STUDY DESIGN:
Intervention Model Description: The intervention group will treated postoperative analgesia with 600 mg of gabapentin plus 65 mcg/kg/hour during 24 hours of nefopam
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GAPA (Experimental): Participants will treated with preoperative 600 mg of gabapentin plus nefopam which will continuously transfused during intraoperative and postoperative 24 hours, and morphine-PCA during postoperative 24 hours
  Interventions: Drug: Gabapentin
- Non-GAPA (No Intervention): Participants will treated with nefopam which will continuously transfused during intraoperative and postoperative 24 hours, and morphine-PCA during postoperative 24 hours

INTERVENTIONS:
Drug: Gabapentin — Gabapentin plus nefopam
  Other Names: Nefopam
  Arms: GAPA

SUMMARY:
The acute pain after spinal surgery is serious. The most pain is during 24 hours after surgery. The multimodal therapy is a method which is applied to treat the postoperative pain.

Morphine is main analgesic to treat postoperative pain. However, some the side-effects can occur to patients and there are associate with dosage. So, some analgesics usually combinate with morphine to postoperative analgesia, include gabapentin, celecoxib, ketamine, ...

Nefopam is a central analgesic. There are effect prevent hyperalgesia. The effect of the combination of gabapentin with nefopam to postoperative analgesia in spinal surgery hasn't been reported yet.

The gabapentin oral with 600 mg combine with continuously intravenous nefopam with 65 µg/kg/hour during 24 hours after spinal surgery whether to increase the effect of postoperative analgesia.

The investigators hypothesized that the gabapentin oral with 600 mg combine with continuously intravenous nefopam with 65 µg/kg/hour during 24 hours after spinal surgery can decrease 40% of the consumption of morphine during 24 hours.

DETAILED DESCRIPTION:
After enrolled, all participants will randomly assigned into the two groups. The intervention group (GAPA-group) will treated preoperative oral 600 mg of gabapentin. After general anesthesia, all participants of both groups will continuously transfused 65 µg/kg/hour of nefopam during 24 hours. After surgery, all cases will treated analgesia with morphine-PCA (2 mg of singe dose, 5 minutes of lockout time, and 6 mg of one hour).

The efficacy of postoperative analgesia will evaluated with the consumption of morphine during 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70.
* Spinal selective surgery

Exclusion Criteria:

* Allergy one of drugs in study.
* Neurological disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Consumption of morphine | Postoperative 24 hours
  Concentration of morphine that participant use during postoperative 24 hours with PCA (mg)

SECONDARY OUTCOMES:
Side-effect | Postoperative 24 hours
  The rate of side-effect induced gabapentin, nefopam, and morphine

CONTACTS AND LOCATIONS:
Overall Officials: Binh V. Huynh, Study Chair — Nhan dan Gia Dinh Hospital
Locations (1):
- Binh Huynh, Ho Chi Minh City, Ho Chi Minh, Vietnam